CLINICAL TRIAL: NCT02484521
Title: Characteristics of Prepulse Inhibition (PPI) of Startle Reflex in Patients With Schizophrenia in Relation to Type of Pharmacological Treatment and Duration of Illness
Brief Title: Prepulse Inhibition (PPI) of Startle Reflex in Schizophrenia Patients Related to Type of Treatment and Illness Duration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Principal Investigator, Elad Haim Kurant, Psychiatry resident, HaEmek Medical Center, Israel
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 0050-15-EMC
Record Dates: First submitted 2015-06-13; First posted 2015-06-29 (Estimated); Last update posted 2020-02-13 (Actual); Status verified 2017-09

CONDITIONS: Inhibition (Psychology); Schizophrenia; Medication Adherence
MeSH Terms: conditions — Inhibition, Psychological; Schizophrenia; Medication Adherence | interventions — Surveys and Questionnaires

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Schizophrenia patients (Active Comparator): Patients diagnosed with Schizophrenia. Will be assigned to PPI monitoring device protocol, according to unified protocol and have questionnaires to assess their status.
  Interventions: Device: PPI monitoring device protocol; Other: Questionnaires
- Healthy subject (Other): This group would be assigned to PPI monitoring device protocol, according to a unified protocol similar to group of patients but not to questionnaires.
  Interventions: Device: PPI monitoring device protocol

INTERVENTIONS:
Device: PPI monitoring device protocol — The investigators would use a monitoring device that would assess startle reflex reaction measured by blinking or the eye. Monitoring would be done with electrodes of EMG device that would be located on orbicularis oculi muscle and will monitor response.
Other: Questionnaires — Group of patients diagnosed with schizophrenia would be interviewed using well validated questionnaires.
  Questionnaires what would be used are:
  1. GAF- Global assessment of functioning
  2. PANSS- Positive and negative syndrome scale
  3. SANS- Scale for the Assessment of Negative Symptoms
  4. The Calgary Depression Scale for schizophrenia
  5. Demographic Questionnaire
  6. Hamilton Anxiety scale
  Arms: Schizophrenia patients

SUMMARY:
PPI is an objective measure to assess pre-attentive processes that have already been tested before in the case of schizophrenia. The investigators aim to assess through this instrument two main characteristics, that the investigators assume are of relevance which are the duration of illness and the type of pharmaceutical treatment, patients receive.

The investigators believe these two main characteristics are critical to the ability of the patients in improvement of their PPI response to startle reflex.

DETAILED DESCRIPTION:
It is common to relate changes of PPI to startle reflex to both negative and positive signs of schizophrenia. Results can both start to explain formations of delusions and hallucinations and the difficulty in processing information for surrounding. It was already tested and discussed in previous trials the relation between type of pharmaceutical treatment as affecting on PPI to startle reflex both causing changes, or improving previous results.

In previous trials as opposed to our planned trial, not much attention was paid for the relation on the changes found to the type of treatment and the duration of the illness. Plus, most trails had different methods of assessing it than our method.

The investigators assume that patients who are receiving typical antipsychotic treatment would have a reduced PPI response to startle reflex compared with those with atypical antipsychotic treatment and those with longer duration of illness would also have reduced PPI response to startle reflex in comparison to those with shorted duration of illness.

The investigators aim to enroll patients already diagnosed with schizophrenia that would be sent by their psychiatrist to the trial. In addition the investigators would enroll control group, not diagnosed with any psychiatric condition.

For both groups, the investigators would run PPI trials according to a unified protocol.

In addition the investigators would run several questionnaires for the group of the patients. Among the details asked of the patient are the duration of the illness and the type of antipsychotic medications they are on and the dosage. Data will then be analyzed.

ELIGIBILITY:
Patients diagnosed with schizophrenia

Inclusion Criteria:

1. Patients diagnosed with schizophrenia or schizoaffective disorder according to Diagnostic and Statistical Manual (DSM) or International Classification of Diseases (ICD).
2. Patients on antipsychotic medications either typical or atypical
3. Patients older than 18 years old and younger than 90 years old
4. In psychiatric follow-up

Exclusion criteria:

1. Patients with earing problems
2. Patients who went through Invasive brain procedure
3. Patients diagnosed with mental retardation
4. Patients with psychoactive substances abuse
5. Pregnant women
6. Patients receiving or received electroconvulsive therapy
7. Patients who have had any medication's regimen changes in either type or dosage in the last month before trial
8. Patients on hormonal therapy

Healthy subjects:

Inclusion criteria:

1. Subjects with no known psychiatric condition
2. Subjects older than 18 years old and younger than 90 years old

Exclusion Criteria:

1. Subjects with earing problems
2. Subjects who went through Invasive brain procedure
3. Subjects diagnosed with mental retardation
4. Subjects with psychoactive substances abuse
5. Pregnant women
6. Subjects on hormonal therapy
7. Subjects with unstable physical status
8. Subjects on psychoactive drug
9. Subjects who have spent time abroad where there is at least 2 hours zone time difference from Israel

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2019-06 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Startle reflex response (anxiety) | 2 hours from arriving to hospital
  Assessed by millivolts registered by electromyography (EMG) electrodes

SECONDARY OUTCOMES:
Prepulse inhibition response (sensorimotor gating) | 2 hours from arriving to the hospital during the time of monitoring
  Assessed by millivolts registered by EMG electrodes
Duration of illness | 4 hours from arriving to the hospital, during questionnaires parts
  Illness duration of longer than 5 years will be considered "long illness duration" while shorter duration than 5 years will be considered "short illness duration" those will then be compared with results of startle and PPI results
Type or class of antipsychotic agents | 4 hours from arriving to the hospital during questionnaires parts
  According to response in demographic questionnaire, a further subdivision of either "Typical" or "Atypical" antipsychotic agent to then be compared with results of startle and PPI results

CONTACTS AND LOCATIONS:
Overall Officials: elad kurante, MD, Principal Investigator — haemek MC
Locations (1):
- Haemek Medical Center, Afula, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Braff DL, Geyer MA, Swerdlow NR. Human studies of prepulse inhibition of startle: normal subjects, patient groups, and pharmacological studies. Psychopharmacology (Berl). 2001 Jul;156(2-3):234-58. doi: 10.1007/s002130100810. PMID 11549226
- [Background] Kohl S, Heekeren K, Klosterkotter J, Kuhn J. Prepulse inhibition in psychiatric disorders--apart from schizophrenia. J Psychiatr Res. 2013 Apr;47(4):445-52. doi: 10.1016/j.jpsychires.2012.11.018. Epub 2013 Jan 1. PMID 23287742
- [Background] Perry W, Minassian A, Feifel D. Prepulse inhibition in patients with non-psychotic major depressive disorder. J Affect Disord. 2004 Aug;81(2):179-84. doi: 10.1016/S0165-0327(03)00157-5. PMID 15306146
- [Background] Geyer MA, Krebs-Thomson K, Braff DL, Swerdlow NR. Pharmacological studies of prepulse inhibition models of sensorimotor gating deficits in schizophrenia: a decade in review. Psychopharmacology (Berl). 2001 Jul;156(2-3):117-54. doi: 10.1007/s002130100811. PMID 11549216
- [Background] Kumari V, Sharma T. Effects of typical and atypical antipsychotics on prepulse inhibition in schizophrenia: a critical evaluation of current evidence and directions for future research. Psychopharmacology (Berl). 2002 Jul;162(2):97-101. doi: 10.1007/s00213-002-1099-x. Epub 2002 Jun 5. PMID 12110987
- [Background] Kishi T, Moriwaki M, Kitajima T, Kawashima K, Okochi T, Fukuo Y, Furukawa O, Naitoh H, Fujita K, Iwata N. Effect of aripiprazole, risperidone, and olanzapine on the acoustic startle response in Japanese chronic schizophrenia. Psychopharmacology (Berl). 2010 Apr;209(2):185-90. doi: 10.1007/s00213-010-1787-x. Epub 2010 Feb 23. PMID 20177883
- [Background] Aggernaes B, Glenthoj BY, Ebdrup BH, Rasmussen H, Lublin H, Oranje B. Sensorimotor gating and habituation in antipsychotic-naive, first-episode schizophrenia patients before and after 6 months' treatment with quetiapine. Int J Neuropsychopharmacol. 2010 Nov;13(10):1383-95. doi: 10.1017/S1461145710000787. Epub 2010 Jul 16. PMID 20633319
- [Background] Swerdlow NR, Light GA, Cadenhead KS, Sprock J, Hsieh MH, Braff DL. Startle gating deficits in a large cohort of patients with schizophrenia: relationship to medications, symptoms, neurocognition, and level of function. Arch Gen Psychiatry. 2006 Dec;63(12):1325-35. doi: 10.1001/archpsyc.63.12.1325. PMID 17146007
- [Background] Csomor PA, Preller KH, Geyer MA, Studerus E, Huber T, Vollenweider FX. Influence of aripiprazole, risperidone, and amisulpride on sensory and sensorimotor gating in healthy 'low and high gating' humans and relation to psychometry. Neuropsychopharmacology. 2014 Sep;39(10):2485-96. doi: 10.1038/npp.2014.102. Epub 2014 May 7. PMID 24801767